CLINICAL TRIAL: NCT01999049
Title: Observational Study of the Argus® II Retinal Prosthesis System
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Foundation Fighting Blindness (Other)
Responsible Party: Sponsor
Other Study IDs: 50813
Record Dates: First submitted 2013-11-25; First posted 2013-12-03 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Argus II Retinal Implant is a revolutionary new device, which offers vision to patients who are blind from retinal degeneration - retinitis pigmentosa. These patients have no alternatives. Patients typically can achieve ambulatory vision.

DETAILED DESCRIPTION:
This study is an investigator-sponsored, observational, controlled, prospective, single-center study. The purpose of this current study is how it affects people's visual function and activities of daily living and to collect additional data on Argus II users in order to monitor the System's safety. In addition, data about the long-term reliability of the System will be gathered.

The Argus II retinal implant will be surgical implanted into patients who are blind but the surgical procedure is not a part of this observational study. Our hypothesis is that the visual results in our hands will be comparable to those reported in the FDA study. We will use the results of this study to plan future enhancements to the service and to explore the use of the device for other blinding conditions.

ELIGIBILITY:
Inclusion Criteria:

•Adults, age 25 years or older with severe to profound outer retinal degeneration.

but some residual light perception. If no residual light perception remains, the retina must be able to respond to electrical stimulation and previous history of useful form vision.

Exclusion Criteria:

* Ocular diseases or conditions that could prevent the Argus II System from working (e.g. optic nerve disease, central retinal artery or vein occlusion, history of retinal detachment, trauma, severe strabismus).
* Ocular structures or conditions that could prevent the successful implantation of the Argus II Implant or adequate healing from surgery (e.g. extremely thin conjunctiva, axial length <20.5 mm or > 26 mm, corneal ulcers, choroidal neovascularisation in the area of the intended tack location, etc.).
* Ocular diseases or conditions (other than cataracts) that prevent adequate visualisation of the inner structures of the eye (e.g. corneal opacity, etc.).
* Inability to tolerate general anaesthesia or the recommended antibiotic and steroid regimen associated with the implantation surgery.
* Predisposition to eye rubbing.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe to profound outer retinal degeneration
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Safety | Patients will be observed for 1 year post-implant.
  The primary endpoint in the study is safety. Safety will be assessed by calculating the proportion of subjects who experience individual procedure- and device-related adverse events. In addition, the proportion of subjects who experience a significant ocular event will also be reported.

SECONDARY OUTCOMES:
Visual function | 1 year
  * Visual function: Visual function means how the eye works (e.g. visual acuity). Visual function will be measured using the following tests: Square Localization; Direction of Motion; Grating Visual Acuity (GVA).
  * Functional vision: Functional vision means how subjects perform in vision-related activities of daily living. Function vision will be assessed using the Functional Low-Vision Observer Rated Assessment (FLORA). A utilization questionnaire will also be administered to track how subjects are using the Argus II System.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Devenyi, MD, Principal Investigator — University Health Network- Toronto Western Hospital
Locations (1):
- UHN Toronto Western Hospital 6E-438, Toronto, Ontario, Canada

REFERENCES:
- [Background] Humayun MS, Dorn JD, da Cruz L, Dagnelie G, Sahel JA, Stanga PE, Cideciyan AV, Duncan JL, Eliott D, Filley E, Ho AC, Santos A, Safran AB, Arditi A, Del Priore LV, Greenberg RJ; Argus II Study Group. Interim results from the international trial of Second Sight's visual prosthesis. Ophthalmology. 2012 Apr;119(4):779-88. doi: 10.1016/j.ophtha.2011.09.028. Epub 2012 Jan 11. PMID 22244176
- [Background] Ahuja AK, Yeoh J, Dorn JD, Caspi A, Wuyyuru V, McMahon MJ, Humayun MS, Greenberg RJ, Dacruz L. Factors Affecting Perceptual Threshold in Argus II Retinal Prosthesis Subjects. Transl Vis Sci Technol. 2013 Apr;2(4):1. doi: 10.1167/tvst.2.4.1. Epub 2013 Apr 12. PMID 24049718